CLINICAL TRIAL: NCT03549247
Title: Evaluation of the Effect of Periodontal Status and Oral Health Consciousness Level on Oral Health Quality of Life by Using OHIP-14 Scale.
Brief Title: Oral Health Related Quality of Life and Periodontal Diseases
Status: Completed | Type: Observational
Sponsor: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, muge lutfioglu, associate professor, Ondokuz Mayıs University
Other Study IDs: OMU KAEK 2015/414
Record Dates: First submitted 2018-04-05; First posted 2018-06-07 (Actual); Last update posted 2018-06-07 (Actual); Status verified 2018-06

CONDITIONS: Periodontal Diseases
Keywords: OHIP-14; Periodontitis
MeSH Terms: conditions — Periodontal Diseases; Periodontitis | interventions — Quality of Life

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- quality of life in periodontal healthy: 250 individuals who have teeth pocket depth is at most 3 mm and there is no loss of attachment, no radiological bone loss and no gingival inflammation determeined for their quality of life
  Interventions: Behavioral: quality of life in healthy,gingivitis,periodontitis groups
- quality of life in gingivitis: 250 individuals who have teeth pocket depth in the mouth is at most 3 mm and there is no loss of attachment, no radiological bone loss and have chronic gingival inflammation with the sign of bleeding determeined for their quality of life
  Interventions: Behavioral: quality of life in healthy,gingivitis,periodontitis groups
- quality of life in periodontitis: 250 individuals who have more than 30% of teeth in the mouth which have pocket depths equal or more than 4mm and clinical attachment levels equal or more than 5mm and have radiologically detected bone loss determeined for their quality of life
  Interventions: Behavioral: quality of life in healthy,gingivitis,periodontitis groups

INTERVENTIONS:
Behavioral: quality of life in healthy,gingivitis,periodontitis groups — a questionnaire form evaluating oral hygiene habits and oral hygiene consciousness levels, OHIP-14 scale was applied

SUMMARY:
The aim of our study was to evaluate the periodontal healthy and diseased individuals with questionnaire, 0ral health impact profile-14(OHIP-14) and dental hygiene fear scale (DHFS) scales and to examine the effect of periodontal disease on the quality of life in relation to oral health consciousness level and fear level against dentist and treatment.

DETAILED DESCRIPTION:
In clinical practice, assessments may provide to detect the disease effected oral sites and the extend of the disease by determining 'objective' surrogate markers but in generally patient based 'subjective' outcomes of those surrogate markers is not evaluated . Oral Health Impact Profile-14 (OHIP-14) is a kind of measurement that is designed to provide a comprehensive detection of the dysfunction,discomfort and disability attributed to oral conditions. Although there are some researchers who have investigated the relationships between patient perceptions and periodontal disease and treatment, further studies are needed to produce more reliable outcomes. It is also well known that psychological and socio demographic status strongly affect the quality of life and these basic key factors of life were also modify the periodontal status of individuals. However, the psychological and socio demographic factors over looked in many of the previous studies,large scale group studies with the survey of quality of life and periodontal status screening are not sufficient. Therefore, the aim of this study was to evaluate the patients with different periodontal status with OHIP-14 scale and a questionnaire to detect the oral health consciousness level.

The protocol of this randomized controlled clinical survey study was approved by the Ethical Committee of the Faculty of Dentistry, ondokuz mayıs university, Turkey, and the study was conducted in accordance with the Declaration of Helsinki. Informed written consent was obtained from all subjects after the details of the clinical procedures were explained. Systematically healthy 750 individuals (subject) aged ≥18 years that referred to the Department of Periodontology, Faculty of Dentistry, ondokuz mayıs University, either for dental treatment or only for dental check-up were included in the study. Prior to dental examination the questionnaire form to detect oral hygiene habits and oral hygiene consciousness levels and the OHIP-14 form to evaluate impact of periodontal status on quality of life were applied to each participants.

Periodontal disease status was determined according to clinical and radiographic criteria. In order to determine the periodontal status of the plaque index(PI), gingival index(GI), probing pocket depth(PPD) and clinical attachment level(CAL) were recorded. Study participants were distributed into three groups as periodontally healthy(H; n=250), gingivitis (G; n=250)and chronic periodontitis (CP; n=250). The relationship between periodontal status with quality of life and perception of how oral health influences the quality of life as well as percieved oral health and oral hygiene consciousness level were evaluted.

Demograhic assesments:

The age, sex, years of education, monthly income, smoking status, oral hygiene habitsvof each participant was recorded.

Assessment of OHIP:

The relationship between periodontal status with quality of life is evaluated with OHIP-14 scale. The validity and reliability of OHIP, consisting of 49 questions, was made by Slade and Spencer . The short form of OHIP was developed due to answering and scoring scales can take a long time and the validity and reliability of OHIP-14 is confirmed by Slade (Slade, 1997). The answers are scored according to the Likert scale. Responses to the items were recorded on a six-point scale: never=0,seldom=1, sometimes=2, fairly often=3, very often=4 and all time=5. The high scores revealed the adversely affected quality of life. The participants were informed on how to complete the indexes. Cronbach's alpha value, which indicates the internal consistency of the scale, is 0.94. The reliability and validity of the Turkish version of the OHIP-14 scale was determined by Mumcu et al. (2006) report.

Assesment of percieved oral health and oral hygiene consciousness level:

The patient based explanation of the periodontal status and the conciousness level and application of oral hygiene measures were detected by applying a questionnaire form.

ELIGIBILITY:
Inclusion Criteria:

* be literate
* systemic healthy
* do not use medication for any reason
* no chemotherapy / radiotherapy story
* not pregnant or in lactation

Exclusion Criteria:

* don't be literate
* have any systemic disease
* use any medication
* chemotherapy/ radiotherapy story
* pregnancy or in lactation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: in our study Ondokuz Mayıs University Faculty of Dentistry Periodontology Clinic evaluated individuals who applied for control and treatment purposes
Sampling Method: Non-Probability Sample
Enrollment: 750 (Actual)
Dates: Start 2015-11-11 (Actual); Primary Completion 2017-07-30 (Actual); Study Completion 2017-10-27 (Actual)

PRIMARY OUTCOMES:
OHIP score to evaluate the oral health related quality of life | 1 day (on the day of examination)
  The changes in OHIP-14 scores (ranging between 0 to 56) determined by the questionnaire applied to the study groups. This questionnare reflected the quality of of life of individual that has oral health problem and the high scores revealed the adversely affected quality of life.
gingival index score for determining periodontal status | 1 day (on the day of examination)
  the gingival index score (ranging 0 to 3) used to define the severity gingival inflammation in order to define the periodontal status.
clinical attachment level measurement for determining periodontal status | 1 day (on the day of examination)
  milimetric measurment of clinical attachement level by using periodontal probe to define the periodontal status.

SECONDARY OUTCOMES:
ages | 1 day (on the day of examination)
  Comparison of ages of healthy, gingivitis and periodontitis groups
marital status | 1 day(on the day of examination)
  Comparison of marital status of healthy, gingivitis and periodontitis groups
education status | 1 day(on the day of examination)
  Comparison of educational status of healthy, gingivitis and periodontitis groups detemined by the duration of education as years
monthly income | 1 day(on the day of examination)
  Comparison of the monthly income of healthy, gingivitis and periodontitis groups detremined by recording the participants as Less than minimum wage, minimum wage, more than minimum wage.
dental visit frequencies | 1 day(on the day of examination)
  Comparison of dental visit frequencies of healthy, gingivitis and periodontitis groups by recording the frequency as when having complaints,sometimes and regularly.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Besiroglu E, Lutfioglu M. Relations between periodontal status, oral health-related quality of life and perceived oral health and oral health consciousness levels in a Turkish population. Int J Dent Hyg. 2020 Aug;18(3):251-260. doi: 10.1111/idh.12443. Epub 2020 May 20. PMID 32367616

DOCUMENTS (1):
  • Study Protocol (2015-10-15): https://cdn.clinicaltrials.gov/large-docs/47/NCT03549247/Prot_000.pdf